CLINICAL TRIAL: NCT02818491
Title: Dexamethasone as an Adjuvant to Ropivacaine for the Interscalene Brachial Plexus Block: a Dose-finding Study
Brief Title: Dexamethasone as an Adjuvant to Ropivacaine for the Interscalene Brachial Plexus Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Eric Albrecht, PD MD, Program director of regional anaesthesia, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CER 217/15
Record Dates: First submitted 2016-06-23; First posted 2016-06-29 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control group (Placebo Comparator): Patients will receive ropivacaine 0.5% 20 mls with normal saline 0.9% 2 mls
  Interventions: Drug: Placebo; Drug: Ropivacaine 0.5%
- Dex 1 (Active Comparator): Patients will receive ropivacaine 0.5% 20 mls with dexamethasone 1 mg in 2 mls
  Interventions: Drug: Dexamethasone 1 mg; Drug: Ropivacaine 0.5%
- Dex 2 (Active Comparator): Patients will receive ropivacaine 0.5% 20 mls with dexamethasone 2 mg in 2 mls
  Interventions: Drug: Dexamethasone 2 mg; Drug: Ropivacaine 0.5%
- Dex 3 (Active Comparator): Patients will receive ropivacaine 0.5% 20 mls with dexamethasone 3 mg in 2 mls
  Interventions: Drug: Dexamethasone 3 mg; Drug: Ropivacaine 0.5%
- Dex 4 (Active Comparator): Patients will receive ropivacaine 0.5% 20 mls with dexamethasone 4 mg in 2 mls
  Interventions: Drug: Dexamethasone 4 mg; Drug: Ropivacaine 0.5%

INTERVENTIONS:
Drug: Placebo — Normal saline 0.9% in 2 mls
  Arms: Control group
Drug: Dexamethasone 1 mg — Dexamethasone 1 mg in 2 mls
  Arms: Dex 1
Drug: Dexamethasone 2 mg — Dexamethasone 2 mg in 2 mls
  Arms: Dex 2
Drug: Dexamethasone 3 mg — Dexamethasone 3 mg in 2 mls
  Arms: Dex 3
Drug: Dexamethasone 4 mg — Dexamethasone 4 mg in 2 mls
  Arms: Dex 4
Drug: Ropivacaine 0.5% — Ropivacaine 0.5% 20 mls

SUMMARY:
Shoulder surgery is associated with moderate to severe postoperative pain. Interscalene brachial plexus block is considered by many as the gold standard for treating postoperative pain and consists of injecting local anaesthetics close to the nerves of the brachial plexus in the neck. Duration of analgesia is between eight to twelve hours depending on the type of administered drugs. Dexamethasone 4 mg is a steroid routinely injected intravenously in anaesthesia for the prophylaxis of postoperative nausea and vomiting. Recently, different trials have demonstrated that combining 4 to 8 mg of dexamethasone with local anaesthetics for a perineural injection may prolong the duration of analgesia up to 24 hours. In a meta-analysis including 29 trials and 1695 patients, investigators have recently demonstrated through a meta-regression that a dose of 4 mg is sufficient and represents a ceiling dose, without neurological complications. The objective of this multicenter randomised controlled double-blinded trial is to determine the optimal dose of perineural dexamethasone. For that purpose, investigators will include a total of 150 patients divided in 5 groups: local anaesthetics with placebo, or with dexamethasone 1, 2, 3 and 4 mg.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for elective shoulder arthroscopy
* duration of surgery less than 4 hours

Exclusion Criteria:

* allergy to local anaesthetics
* history of neck surgery
* history of neck radiotherapy
* severe respiratory disease
* diabetic patient
* chronic pain condition
* pregnancy
* patient suffering from cancer
* patient with addicted disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Duration of analgesia | 24hour

SECONDARY OUTCOMES:
Duration of motor block | 24hour
Onset time of action of sensory block | 1hour
Onset time of action of motor block | 1hour
Equivalent morphine consumption in postanesthetic care unit | 4hour
Equivalent morphine consumption on postoperative day 1 | 24hour
Pain scores at rest in postanesthetic care unit (visual analogue scale, 0-10) | 4hour
Pain scores on movement in postanesthetic care unit (visual analogue scale, 0-10) | 4hour
Pain scores at rest on postoperative day 1 (visual analogue scale, 0-10) | 24hour
Pain scores on movement on postoperative day 1 (visual analogue scale, 0-10) | 24hour
Rate of postoperative nausea and vomiting (PONV) | 24hour
  Presence of PONV (YES/NO)
Rate of pruritus | 24hour
  Presence of pruritus (YES/NO)
Satisfaction score on postoperative day 1 (visual analogue scale, 0-10) | 24hour
Glycemia in postanesthetic care unit (mmol/l) | 4hour
Rate of infection | 24hour
  Presence of infection (YES/NO)
Rate of infection | 7 days
  Presence of infection (YES/NO)
Rate of paresthesia | 7 days
  Presence of paresthesia (YES/NO)
Rate of muscle weakness | 7 days
  Presence of muscle weakness (YES/NO)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Albrecht, MD, Study Director — Centre Hospitalier Universitaire Vaudois; Matthias Matthias, MD, Principal Investigator — AZ Groeninge Hospital, Pres. Kennedylaan 4, 8500 Kortrijk, Belgium
Locations (1):
- AZ Groeninge Hospital, Kortrijk, Belgium

IPD SHARING:
Plan to Share IPD: Undecided